CLINICAL TRIAL: NCT02943603
Title: A Phase II Study of Perioperative mFOLFOX6 Chemotherapy Plus Pembrolizumab(MK-3475) Combination in Patients With Potentially Resectable Adenocarcinoma of the Gastroesophageal Junction (GEJ) and Stomach
Brief Title: A Study of Perioperative mFOLFOX6 Plus Pembrolizumab in Patients With Potentially Resectable Adenocarcinoma of the Gastroesophageal Junction (GEJ) and Stomach
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled. PI/Sponsor left UPitt. IND withdrawn & revised protocol submitted through the new institution. New study recruiting under NCT03488667.
Sponsor: Weijing Sun, MD, FACP (Other)
Responsible Party: Sponsor-Investigator, Weijing Sun, MD, FACP, Professor of Medicine, University of Pittsburgh School of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-104
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2017-09

CONDITIONS: Adenocarcinoma; Stomach Cancer
Keywords: mFOLFOX6; pembrolizumab
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mFOLFX6 + Pembrolizumab (Experimental): Subjects will receive mFOLFOX6 every 2 weeks (on Days 1, 15, 29, 43) and Pembrolizumab every 3 weeks (on Days 1, 22, 43).
  Interventions: Drug: mFLOFOX6 + pembrolizumab

INTERVENTIONS:
Drug: mFLOFOX6 + pembrolizumab — the combination of mFOLFOX6 + pembrolizumab is the single intervention even though the is dosed differently.

SUMMARY:
This research study is being down to find what, effects, good and/or bad, adding Pembrolizumab to standard chemotherapy mFOLFOX before and after surgery have on the patient and the patient's cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically-confirmed diagnosis of adenocarcinoma of the GEJ or stomach.
* Have newly diagnosed localized or locally advanced (T1N1-3M0 or T2-4NanyM0), potentially resectable disease without any prior systemic chemotherapy.
* Have no evidence of distant metastases (as determined by EUS, PET-CT or staging laparoscopy).
* Be eligible and reasonably fit to undergo potentially curative resection
* Must be 18 - 75 years of age.
* 6. Be willing and able to provide written informed consent/assent for the trial.
* Have measurable disease based on RECIST 1.1.
* Have pre-resection tissue (EGD or EUS biopsy from the diagnosis) available.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function:
* Be willing to provide blood and tissue samples for research purposes
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Has received prior chemotherapy for any malignant disorder, thoracic radiation therapy or prior surgical resection of an esophagogastric tumor.
* Has biopsy-proven invasion of tracheobronchial tree or tracheo-esophageal fistula.
* Has distant metastatic disease on imaging or staging laparoscopy at the time of study entry.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Clinically significant (≥ grade 2) peripheral neuropathy at the time of study entry.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B or Hepatitis C.
* Inoperable on the basis of co-existent medical problems.
* Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude any of the study drugs.
* Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response [ypCR] | Up to 12 weeks
  Number of participants with pathological complete response [pCR] at 12 weeks/total number of evaluable participants.
number of adverse events related to toxicity | up to 18 months for accrual + 12 months of intervention and 1 month of safety follow-up for last subject (31 months)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 weeks
  Number of participants with response (partial response + complete response) at 12 weeks/total number of evaluable participants.
Disease Free Survival post surgery | up to 18 months for accrual + 1 month for screening and 3 months of intervention before surgery for last subject then 12 months of follow-up (34 months)
Overall Survival (OS) | up to 18 months for accrual + 12 months of intervention for last subject (30 months)
PET response | up to 18 months for accrual + 1 month for screening and 3 months of intervention for last subject (22 months)
PD-L1 expression in tumor cells | up to 18 months for accrual + 1 month for screening and 3 months of intervention for last subject (22 months)
  change in PD-L1 expression on the surface and in the nucleus of the tumor cells over treatment will be related to ypCR by means of logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Weijing Sun, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States